CLINICAL TRIAL: NCT01295502
Title: A Phase I Evaluation of Extended Field Radiation Therapy With Concomitant Cisplatin Chemotherapy Followed by Paclitaxel and Carboplatin Chemotherapy in Women With Cervical Carcinoma Metastatic to the Para-aortic Lymph Nodes
Brief Title: Cisplatin and Radiation Therapy Followed by Paclitaxel and Carboplatin in Treating Patients With Stage IB-IVA Cervical Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9926; NCI-2011-02665 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695304; GOG-9926 (Other: NRG Oncology); GOG-9926 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB Cervical Cancer AJCC v6 and v7; Stage IIA Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage IIIA Cervical Cancer AJCC v6 and v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Brachytherapy; Paclitaxel; Taxes

ARMS (1):
- Treatment (radiation, cisplatin, paclitaxel, carboplatin) (Experimental): Patients receive cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36 and undergo extended-field radiotherapy daily 5 days a week for 6 weeks followed by brachytherapy. Beginning 4-6 weeks after completion of chemoradiation, patients receive adjuvant chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Internal Radiation Therapy; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Radiation: Internal Radiation Therapy — Undergo brachytherapy
  Other Names: BRACHYTHERAPY; internal radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase I trial studies the side effects and the best dose of paclitaxel and carboplatin after cisplatin and radiation therapy in treating patients with stage IB-IVA cervical cancer. Drugs used in chemotherapy, such as cisplatin, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving paclitaxel and carboplatin after cisplatin and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) and dose-limiting toxicities (DLT) of adjuvant carboplatin and paclitaxel chemotherapy following concurrent weekly cisplatin chemotherapy and extended field radiation in women with newly diagnosed stage IB-IVA cervical cancer, with positive para-aortic nodes.

II. To determine the feasibility of the treatment regimen over the four cycles of adjuvant chemotherapy once the MTD is estimated.

III. To assess the toxicities of the treatment regimen the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OBJECTIVES:

I. To assess the response rate to this treatment regimen in patients with measurable disease.

II. To examine progression-free survival for one year on this treatment regimen.

III. To examine overall survival. IV. To examine the location of recurrence, loco-regional versus distant for one year after completion of therapy.

V. To estimate the frequency of chronic toxicities experienced within one year of study entry.

OUTLINE: This is a dose-escalation study of carboplatin and paclitaxel.

Patients receive cisplatin intravenously (IV) over 1 hour on days 1, 8, 15, 22, 29, and 36 and undergo extended-field radiotherapy daily 5 days a week for 6 weeks followed by brachytherapy. Beginning 4-6 weeks after completion of chemoradiation, patients receive adjuvant chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed cervical cancer (squamous, adenocarcinoma, or adenosquamous): International Federation of Gynecology and Obstetrics (FIGO) clinical stages IB, IIA, IIB, IIIA, IIIB, IVA, with positive para-aortic lymph nodes confirmed by positron emission tomography (PET)/computed tomography (CT) scan, fine needle biopsy, extraperitoneal biopsy, laparoscopic biopsy or lymphadenectomy
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0-2
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 100,000/mcl
* Creatinine =< institutional upper limit normal (ULN); Note: if creatinine > ULN, creatinine clearance must be > 50 mL/min
* Bilirubin =< 1.5 times ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Neuropathy (sensory and motor) =< grade 1
* Patients with ureteral obstruction must undergo stent or nephrostomy tube placement prior to study entry
* Patients must meet the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients of child-bearing potential must have a negative serum pregnancy test prior to study entry (within 72 hours prior to initiation of study treatment) and be practicing an effective form of contraception; women should not breast-feed while on this study
* Patients must not be receiving any other investigational agent
* Patients should have an audiogram at baseline, and patients with pre-existing hearing loss or hearing loss during treatment should be assessed frequently during cisplatin therapy

Exclusion Criteria:

* Patients who have received previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy
* Patients with active infection
* Patients who have circumstances that will not permit completion of this study or the required follow-up
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have undergone major surgery, excluding diagnostic biopsy, within 30 days (to allow for full recovery) prior to registration
* Patients who have a significant history of cardiac disease, (i.e., uncontrolled hypertension, unstable angina, congestive heart failure, or uncontrolled arrhythmias) within 6 months of registration
* Patients who have a known sensitivity reactions to products containing Cremophor EL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-04-04 (Actual); Primary Completion 2019-12-02 (Estimated)

PRIMARY OUTCOMES:
MTD of adjuvant carboplatin and paclitaxel determined based on the dose-limiting toxicities assessed by NCI CTCAE version 4 | 21 days

SECONDARY OUTCOMES:
Objective tumor response rate in patients enrolled with measurable disease | Up to 1 year
  Will be tabulated overall.
Progression-free survival (PFS) | Time from study entry to time of progression or death, whichever occurs first, assessed at 1 year
  PFS will be summarized using Kaplan-Meier plots.
Overall survival | Time from study entry to time of death or the date of last contact, assessed up to 1 year
  Survival will be summarized using Kaplan-Meier plots.
Location of recurrence (loco-regional versus distant) defined as newly evident disease for patients who have no evidence of disease at baseline or progressive disease for patients who have strictly non-measurable disease at baseline | Up to 1 year
Chronic toxicities experienced classified using the CTCAE version 4 | Within 1 year of study entry

CONTACTS AND LOCATIONS:
Overall Officials: Cecelia H Boardman, Principal Investigator — NRG Oncology
Locations (14):
- United States (14):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Augusta University Medical Center, Augusta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia